CLINICAL TRIAL: NCT05078073
Title: Hyperbaric Oxygen Therapy Improve Acute Graft-Versus-Host Disease in Patients Underwent Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: HBOT in the Treatment and Prevention of aGVHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Head of Depertment of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBOT in aGVHD
Record Dates: First submitted 2021-09-06; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Hyperbaric Oxygen Therapy; Acute-graft-versus-host Disease
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aGVHD-HBOT (Experimental): Patients after allo-HSCT will receive hyperbaric oxygen therapy (HBOT) on the next day of the aGVHD diagnosis was determined.
  Interventions: Device: Hyperbaric oxygen therapy
- aGVHD-HBOT free (No Intervention): Patients after allo-HSCT will NOT receive hyperbaric oxygen therapy (HBOT) on the next day of the aGVHD diagnosis was determined.

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — Patients with aGVHD treated with HBOT every two days
  Arms: aGVHD-HBOT

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative therapeutic strategy for patients with hematopoietic malignancies. However, the therapeutic benefits and wider application of allo-HSCT are limited by acute graft-versus-host disease (aGVHD), the latter remains a major obstacle against long-term survival for this population. New aGVHD prophylactic and therapeutic strategies that are superior in efficacy, safety, cost-effectiveness, and less technically demanding are still in desperate need. Hyperbaric oxygen therapy (HBOT) has been confirmed as an effective and economical therapeutic modality for hemorrhagic cystitis (HC) whether induced by infection or acute graft-versus-host disease (aGVHD) for transplant recipients. However, little is known about its involvement in aGVHD. In this study, the investigators designed a randomized, controlled, and open clinical trial to confirm the safety and efficacy of HBOT on aGVHD in patient underwent allo-HSCT.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative therapeutic strategy for patients with hematopoietic malignancies. However, the therapeutic benefits and wider application of allo-HSCT are limited by acute graft-versus-host disease (aGVHD), the latter remains a major obstacle against long-term survival for this population. New aGVHD prophylactic and therapeutic strategies that are superior in efficacy, safety, cost-effectiveness, and less technically demanding are still in desperate need.

Although a variety of immune and non-immune cells are involved in the development of aGVHD, reactive oxygen species (ROS) has been proved as the primary triggers of the inflammatory response and play a key role in the pathogenesis of aGVHD. Therefore, strategies targeting ROS production are crucial for effectively managing aGVHD. Hyperbaric oxygen therapy (HBOT) is a well-established treatment method, which is used to improve non-healing ulcers secondary to aGVHD and hemorrhagic cystitis (HC) after allo-HSCT whether induced by infection or aGVHD. Even the exact mechanism is not fully understood, HBOT was demonstrated to reduce a series of pro-inflammatory cytokines release and can improve the action of antibiotics.

In this study, the investigators plan to initiate a randomized, controlled, and open clinical cohort study confirm the safety and efficacy of HBOT on aGVHD in patient underwent allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic stem cell transplantation
* Patients develop aGVHD
* The count of neutrophilia cells over 0.5 * 109/L, hemoglobin over 60 g/L, platelet over 30 *109/L
* Signed informed consent

Exclusion Criteria:

* Unsuitable to the study due to severe complication such as uncontrolled severe infection
* Claustrophobia
* Ear diseases such as otitis media
* Eye diseases such as glaucoma
* Epilepsy history
* Important organ dysfunction
* Coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of HBOT as complete response or partial response for the treatment of aGVHD | Four years
  Complete or partial response rate of HBOT for the treatment of aGVHD will be measured using Bayesian method.
Incidence of aGVHD when HBOT was administrated as prophylaxis measurement at one month after transplant | 100 days post transplant
  At one month after transplant, HBOT will be administrated every three days (up to 6 times) to recipients without aGVHD evidence, the incidence of aGVHD will be counted.

SECONDARY OUTCOMES:
Overall survival rate | Four years
  Will be summarized by frequency and 95% confidence interval. The distribution of time-to-event endpoints will be estimated by Kaplan-Meier estimate. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazards regression will be employed for multivariate analysis on time-to-event outcomes.
Leukemia-free survival rate | Four years
  Will be summarized by frequency and 95% confidence interval. The distribution of time-to-event endpoints will be estimated by Kaplan-Meier estimate. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazards regression will be employed for multivariate analysis on time-to-event outcomes.
Relapse rate | Four years
  Relapse rate of recipients will be measured using Bayesian method. Will be summarized by frequency and 95% confidence interval.
Incidence of adverse events of HBOT | Four years
  Toxicities will be summarized by grade and by their relationship to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zhou, Dr., Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No